CLINICAL TRIAL: NCT07212153
Title: The Effect of Preoperative Oral Carbohydrate Loading on Insulin Resistance in Adult Patients Undergoing Cardiac Surgery
Brief Title: Impact of Preoperative Oral Carbohydrate Loading on Insulin Resistance in Adult Cardiac Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rifdhani Fakhrudin Nur (Other)
Responsible Party: Sponsor-Investigator, Rifdhani Fakhrudin Nur, Principal Investigator, Gadjah Mada University
Organization: Gadjah Mada University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: RIF-RCT2025-001
Record Dates: First submitted 2025-09-22; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Cardiac Surgery; Insulin Resistance
Keywords: carbohydrate loading; insulin resistance; cardiac surgery; HOMA-IR
MeSH Terms: conditions — Insulin Resistance | interventions — maltodextrin; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is double-blind. Participants, care providers (surgeons, anesthesiologists, ICU staff), investigators, outcome assessors, data collectors, and analysts were blinded to group allocation. Only the designated study staff who handled randomization and intervention preparation had access to allocation information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbohydrate Loading (CL) (Experimental): Participants receive 400 mL of a maltodextrin-based carbohydrate drink 2 hours before surgery. The drink contains 50 g of carbohydrate (maltodextrin).
  Interventions: Dietary Supplement: Oral Carbohydrate Drink (Maltodextrin)
- Placebo Loading (PL) (Placebo Comparator): Participants receive 400 mL of plain water 2 hours before surgery, following the same timing and fasting protocol as the experimental group.
  Interventions: Other: Placebo (Water)

INTERVENTIONS:
Dietary Supplement: Oral Carbohydrate Drink (Maltodextrin) — Participants receive 400 mL of a clear beverage containing 50 g of maltodextrin (carbohydrate) 2 hours before anesthesia induction. The drink is used to lower insulin resistance and improve perioperative recovery.
  Other Names: Preoperative carbohydrate loading drink
  Arms: Carbohydrate Loading (CL)
Other: Placebo (Water) — Participants receive 400 mL of plain water 2 hours before anesthesia induction, following the same protocol and timing as the carbohydrate drink group.
  Other Names: Clear water placebo
  Arms: Placebo Loading (PL)

SUMMARY:
The goal of this clinical trial is to investigate the effect of preoperative oral carbohydrate on insulin resistance in adult cardiac surgery patients with a cardiopulmonary bypass machine. Insulin resistance is when the body does not respond well to insulin, which can raise blood sugar and slow recovery.

The main question this study aims to answer is:

Does drinking a carbohydrate drink 2 hours before surgery lower insulin resistance compared to drinking only water after on pump cardiac surgery?

Researchers will compare two groups:

One group will drink 400 milliliters of a maltodextrin (carbohydrate) drink (CL group). The other group will drink 400 milliliters of water (PL group).

Participants will:

1. Be randomly assigned to one of the two groups.
2. Have blood samples taken to measure insulin and glucose before and after surgery (at hour-0, and hour-24 after ICU admission).
3. Be monitored in the intensive care unit for 24 hours after surgery.

DETAILED DESCRIPTION:
This prospective, randomized controlled trial is designed to evaluate whether preoperative oral carbohydrate loading reduces perioperative insulin resistance in adults undergoing elective cardiac surgery at Dr. Sardjito Hospital, Yogyakarta, Indonesia. Fifty participants aged 20-60 years with American Society of Anesthesiologists (ASA) physical status II-III will be randomly assigned to one of two groups:

1. Intervention group (Carbohydrate Loading, CL): participants will receive 400 milliliters of a maltodextrin-based carbohydrate drink 2 hours before anesthesia.
2. Control group (Placebo Loading, PL): participants will receive 400 milliliters of plain water 2 hours before anesthesia.

All participants will follow standard preoperative fasting guidelines. Blood samples for glucose and insulin will be taken immediately after induction of anesthesia, upon ICU admission (hour 0), and at hour 24 in the ICU. The main outcome is the Homeostatic Model Assessment of Insulin Resistance (HOMA-IR). Secondary outcomes include perioperative glucose levels and postoperative insulin requirements.

Randomization is computer-generated, with allocation concealed until assignment. Surgeons, anesthesiologists, ICU staff, outcome assessors, and data analysts will be blinded to group allocation. The sample size of 50 participants (25 per group) was calculated based on prior effect sizes, with 80% power and a two-sided alpha of 0.05.

Data will be analyzed using descriptive statistics and appropriate tests for continuous and categorical variables. Between-group comparisons will use Student's t-test or Mann-Whitney U test as appropriate. Normality will be assessed by Shapiro-Wilk test. Repeated measures will be analyzed with paired tests or ANCOVA models. A p-value <0.05 will be considered statistically significant.

This study is expected to provide new evidence on whether preoperative carbohydrate loading can reduce insulin resistance in the specific context of cardiac surgery, and potentially improve perioperative management and patient recovery.

ELIGIBILITY:
Inclusion criteria:

* Age 20 to 60 years
* ASA physical status II or III
* Good tolerance to enteral fluid administration

Exclusion criteria:

* History of diabetes mellitus
* Thyroid insufficiency
* Adrenal insufficiency
* Gastroesophageal reflux disease
* Emergency cardiac surgery

Dropout criteria:

* Participant withdraws consent
* Cardiac surgery duration exceeds 4 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
HOMA-IR (Homeostasis Model Assessment for Insulin Resistance) | baseline, 0 hour ICU admission, and 24 hours ICU admission
  The Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) is calculated as fasting insulin (µU/mL) × fasting glucose (mmol/L) / 22.5. Higher values indicate greater insulin resistance.

SECONDARY OUTCOMES:
Perioperative Blood Glucose Levels | baseline, 0 hour ICU admission, and 24 hours ICU admission
  Blood glucose measured from central venous samples to assess changes in glucose metabolism during and after cardiac surgery.
Perioperative Serum Insulin Concentration | baseline, 0 hour ICU admission, and 24 hours ICU admission
  Serum insulin level measured from central venous blood samples to characterize perioperative insulin changes. Higher values indicate higher circulating insulin.

CONTACTS AND LOCATIONS:
Locations (1):
- RSUP Dr. Sardjito, Sleman, D.I.Yogyakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be made available upon reasonable request to the corresponding investigator after publication of study results.
Supporting Information: Study Protocol, SAP, ICF